CLINICAL TRIAL: NCT07041034
Title: The Effectiveness of the Systematic Unmet Needs Assessment and Management (SUNAM) Protocol on Behavioral and Psychological Symptoms of Institutionalized Residents With Dementia
Brief Title: SUNAM Protocol for Managing BPSD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mackay Medical College (Other)
Responsible Party: Principal Investigator, Chin-Tsung Shen, The Office of Research and Development, Mackay Medical College
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MMC-RD-113-1B-P016
Record Dates: First submitted 2025-06-19; First posted 2025-06-27 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-05

CONDITIONS: Behavioral and Psychological Symptoms of Dementia
Keywords: Virtual Reality, SUNAM Protocol, Dementia Care, Behavioral and Psychological Symptoms (BPSD), Caregiver Training, Unmet Needs
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): This group will receive BPSD foundational education, VR-based training and SUNAM protocol.
  Interventions: Behavioral: Experimental Group
- Active Comparator Group (Active Comparator): This group will receive BPSD foundational education and VR-based training.
  Interventions: Behavioral: Active Comparator Group

INTERVENTIONS:
Behavioral: Active Comparator Group — The group will receive:
  1.Foundational Education: A structured session introducing key concepts of BPSD, symptom recognition, and general management approaches. 2.Simulation-Based Training: An interactive training module using case-based simulation to illustrate common BPSD scenarios and guide caregivers in applying appropriate strategies.
  This group will not receive the protocol-based intervention component.
  Arms: Active Comparator Group
Behavioral: Experimental Group — The intervention consists of three components:
  1. Foundational Education: A structured session introducing key concepts of BPSD, symptom recognition, and general management approaches.
  2. Simulation-Based Training: An interactive training module using case-based simulation to illustrate common BPSD scenarios and guide caregivers in applying appropriate strategies.
  3. SUNAM Protocol Training: Instruction on a structured, theory-informed protocol aimed at identifying and addressing underlying factors that contribute to BPSD in institutionalized residents.
  Arms: Experimental Group

SUMMARY:
This study evaluates the effectiveness of the Systematic Unmet Needs Assessment and Management (SUNAM) Protocol, an algorithm-based intervention developed from the unmet needs theory of BPSD, in reducing Behavioral and Psychological Symptoms of Dementia (BPSD) among institutionalized residents. Both the experimental and control groups received 100 minutes of BPSD foundational education and 100 minutes of VR simulation training. The experimental group received an additional 150 minutes of SUNAM protocol training. The study aims to determine whether integrating SUNAM into caregiver training enhances BPSD assessment, management, and reduction by addressing unmet needs.

DETAILED DESCRIPTION:
Background:Behavioral and Psychological Symptoms of Dementia (BPSD) are common and distressing for dementia residents and their caregivers. These symptoms often arise from unmet needs, yet current care practices frequently fail to systematically identify and address them. As a result, effective management of BPSD remains a significant challenge in long-term care settings.

Purpose:This study aims to evaluate the effectiveness of the Systematic Unmet Needs Assessment and Management (SUNAM) Protocol, an algorithm-based intervention developed based on the unmet needs theory of BPSD. The intervention focuses on identifying and addressing unmet needs to reduce BPSD and improve care outcomes by enhancing caregivers' ability to manage these symptoms more effectively.

Methods:This is a cluster-randomized controlled trial with a repeated measures design conducted across long-term care (LTC) facilities. Both the experimental and control groups received 100 minutes of BPSD foundational education and 100 minutes of VR-based training. The experimental group additionally received 150 minutes of training on the Systematic Unmet Needs Assessment and Management (SUNAM) Protocol, an algorithm-based intervention developed to identify and address unmet needs related to BPSD. Resident data, including demographics, medical conditions, Barthel Index, and MMSE scores, were collected. Outcome measures included the frequency of BPSD, the number of unmet needs, and the frequency of BPSD assessment and management, all of which were assessed for the past two weeks at three time points (pre-intervention, two weeks after the intervention, and four-week follow-up). Data analysis was performed using SPSS 25.0, with descriptive statistics and mixed linear models to examine improvements within and between groups over time.

ELIGIBILITY:
Inclusion Criteria:

* a. Diagnosed with dementia or documented as having dementia in medical records. b. Currently residing in the long-term care facility.

Exclusion Criteria:

* a. Diagnosed with schizophrenia. b. Residents whose legal representative does not provide consent for participation.

Ages: 65 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-06-28 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of BPSD assessment and management. | Baseline, 2-week post-intervention, and 4-week follow-up.
  Measured using a structured checklist documenting the weekly frequency (over the past two weeks) of caregivers' assessment of BPSD, use of non-pharmacological interventions, and referrals to other professionals.
Change in number of unmet needs. | Baseline, 2-week post-intervention, and 4-week follow-up.
  Measured using a 27-item Dementia Unmet Needs Checklist covering physical, psychological, social, and environmental domains. Items are rated yes/no (1/0), with higher scores indicating more unmet needs.

SECONDARY OUTCOMES:
Change in frequency of BPSD symptoms. | Baseline, 2-week post-intervention, and 4-week follow-up.
  Measured using a 34-item composite checklist developed by integrating the 29 items from the Cohen-Mansfield Agitation Inventory (CMAI) with five additional commonly observed emotional and psychiatric symptoms in dementia (e.g., anxiety, depression, hallucinations, delusions, refusal to eat or care), with each item rated on a 7-point scale based on observed frequency over the past two weeks. Higher scores reflect greater symptom severity.

IPD SHARING:
Plan to Share IPD: No